CLINICAL TRIAL: NCT01975012
Title: A Phase I/II, Open-Label Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Rilpivirine in Antiretroviral Naive HIV-1 Infected Children, < 12 Years of Age
Brief Title: Safety, Tolerability, Drug Interactions, and Antiviral Activity of Rilpivirine in Antiretroviral-Naive HIV-Infected Children Less Than 12 Years of Age
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1111; 11902 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: 6 to less than 12 years of age (Experimental): Participants in this arm will be at least 6 but younger than 12 years of age; they will receive the study drug RPV together with 2 other NRTIs.
  Interventions: Drug: Rilpivirine
- Cohort 2: 2 to less than 6 years of age (Experimental): Participants in this arm will be at least 2 but younger than 6 years of age; they will receive the study drug RPV together with 2 other NRTIs.
  Interventions: Drug: Rilpivirine

INTERVENTIONS:
Drug: Rilpivirine — For Cohort 1, Stage 1: RPV will be given orally as a 25-mg film-coated tablet (or for dosing in younger children, as granules [2.5 mg/g]) each day with a meal.
  For Cohort 1, Stage 2: The dose of RPV will be determined once Cohort 1, Stage 1 data are available.
  For Cohort 2: The dose of RPV will be determined once Cohort 1 data are available.
  Other Names: RPV, TMC278, Edurant

SUMMARY:
Development of tolerable and effective antiretroviral (ARV) drugs for use in children and adolescents remains a high priority. First-line therapy with non-nucleoside reverse transcriptase inhibitors (NNRTIs) has proven to be effective for HIV-1-infected infants, children, and adolescents. This study will evaluate the safety, effectiveness, and dosing levels of the NNRTI rilpivirine (RPV) when given with two other ARV drugs in treatment-naive, HIV-1-infected children less than 12 years of age.

DETAILED DESCRIPTION:
This study will enroll HIV-1-infected children less than 12 years of age who are naive to antiretroviral therapy (ART) (have never taken ARV drugs). Study participants will be assigned to 1 of 2 cohorts based on age. Cohort 1 will include children at least 6 years of age to less than 12 years of age. Cohort 2 will include children at least 2 years of age to less than 6 years of age. Each cohort will consist of two stages: Stage 1 and Stage 2. Stage 1 will be the initial dose finding stage. Participants will begin treatment with daily RPV and 2 nucleoside reverse transcriptase inhibitors (NRTIs). The 2 NRTIs will be selected by the site investigator but will not be provided through the study. This stage of the study will involve intense pharmacokinetic (PK) sampling to evaluate the safety, tolerability, and antiviral activity of RPV, which will allow for the selection of an RPV dose to use in Stage 2 of the study. Participants in both cohorts will remain on RPV-based therapy for up to 48 weeks.

Study enrollment will begin with Cohort 1. Once data from Cohort 1 has been reviewed and an RPV dose has been approved, enrollment for Cohort 2 will begin.

Study participation will include at least 12 study visits over 48 weeks. Participants who complete 48 weeks of RPV treatment and are benefiting from the drug will continue on the study and receive RPV as part of a long-term safety follow-up for a minimum of 4 additional years. Study visits in this stage of the study will occur every 24 weeks.

At most visits, participants will give a medical history and undergo a physical exam, blood collection, and urine collection. At some visits, participants will also undergo an electrocardiogram (ECG), adrenocorticotropic hormone (ACTH) stimulation test (consisting of blood collection and an injection of ACTH), and determination of the participant's stage of sexual development.

ELIGIBILITY:
Inclusion Criteria - Stage 1, Step 1 and Stage 2

* A confirmed HIV-1 infection. More information on this criterion can be found in the protocol.
* Participant has never been treated with an HIV vaccine
* No evidence of prior ARV drug use with the exception of prior use of zidovudine (AZT) for up to 6 weeks to prevent mother-to-child transmission
* HIV-1 plasma viral load (VL) at screening greater than 500 HIV-1 RNA copies/mL but less than or equal to 100,000 HIV-1 RNA copies/mL (assayed by RNA polymerase chain reaction [PCR] standard specimen procedure) Note: Participants may be re-screened once only, if their baseline VL does not meet the entry criteria.
* In the judgment of the investigator, it is appropriate to initiate ARV therapy based on the participant's medical condition and taking into account guidelines for the treatment of HIV-1 infection in children
* Results from the genotypic resistance testing at screening demonstrate sensitivity to the selected NRTIs for the chosen background regimen
* Able to swallow whole tablets (Cohort 1 initial dose only)
* Female participants who are of childbearing potential and who are engaging in sexual activity that could lead to pregnancy, must use two adequate birth control methods while on study and for 4 weeks after stopping study drug. More information on this criterion can be found in the protocol.

Inclusion Criteria - Stage 1, Step 2

* Participants belonging to a cohort that failed Stage 1 Step 1 initial dose that meet the following criteria (as determined by the study team): Are able to have an adjustment in study drug dose (and the new dose would not exceed 25 mg) and appear to have room to stay within therapeutic range on the new dose

Exclusion Criteria - Stage 1, Step 1 and Stage 2

* Having documented genotypic evidence of RPV resistance. More information on this criterion can be found in the protocol.
* Documented evidence of infection during breastfeeding by a mother taking NNRTI-based ART. If there are no data or no history available then the participant would be eligible as long as all other inclusion and exclusion criteria are fulfilled.
* Documented evidence of maternal NNRTI use during pregnancy. If there are no data or no history available then the participant would be eligible as long as all other inclusion and exclusion criteria are fulfilled.
* Previously documented HIV-2 infection in participant or participant's mother. If there are no data or no history available then the participant would be eligible as long as all other inclusion and exclusion criteria are fulfilled.
* Use of disallowed medication from 4 weeks prior to the entry visit or anticipated use of any disallowed medications
* A) Participant has used chronic systemic immunosuppressive agents within 30 days prior to entry or is anticipated to need chronic systemic immunosuppressive agents during the study. Short courses of systemic corticosteroids (e.g., prednisone or equivalent up to 2 mg/kg/day for less than or equal to 7 days) are permitted, as long as the use was greater than 30 days prior to entry; B) participant has used both chronic inhaled and intranasal steroids within 30 days prior to entry. Use of either inhaled or intranasal steroids are allowed.
* Participant has any active AIDS-defining illness (Category C conditions according to the Centers for Disease Control and Prevention [CDC] revised Classification System for HIV Infection 1994), within 30 days prior to screening. Stable not currently active conditions that are not likely to interfere with safety assessments may be allowed with permission from the protocol team.
* Any active clinically significant disease or findings (other than HIV infection) during screening or medical history or physical examination that in the investigator's opinion, would compromise the outcome of the study
* Any confirmed Grade 3 or 4 laboratory toxicity according to the Division of AIDS (DAIDS) grading table at screening, except for: asymptomatic Grade 3 absolute neutrophil count decrease; asymptomatic Grade 3 platelet count decrease; asymptomatic Grade 3 total amylase, triglyceride, cholesterol elevation
* Participant has active tuberculosis and/or is being treated for tuberculosis at screening
* Participant has one or more of the following risk factors for ECG QTc prolongation:

  * A confirmed prolongation of QT/QTc interval, (e.g., repeated demonstration of QTcF [Fridericia correction] interval greater than 450 ms in the screening ECG (i.e., retesting to reassess eligibility will be allowed once using an unscheduled visit during the screening period)
  * Pathological Q-waves (defined as Q-wave greater than 40 ms or depth greater than 0.4-0.5 mV)
  * Evidence of ventricular pre-excitation
  * Electrocardiographic evidence of complete right or complete or incomplete left bundle branch block
  * Evidence of second or third degree heart block
  * Intraventricular conduction delay with QRS duration greater than 120 ms
  * Bradycardia as defined by sinus rate less than 50 bpm
  * Personal or family history of long QT syndrome
  * Personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, with the exception of sinus arrhythmia
  * Syncopal episodes
  * Risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia)
* Participant's family is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate to a non-IMPAACT study site during the study
* Hepatitis B virus surface antigen (HBsAg) positive or hepatitis C virus (HCV) antibody positive
* Any history of malignancy
* Participant enrolled in another clinical trial of an investigational agent or experimental vaccine or a compound or device which is not commercially available
* Any history of adrenal insufficiency
* Pregnancy or breastfeeding if of childbearing potential

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Failure to meet PK guidelines | Measured through Week 48
  Main PK parameters include the area under the plasma concentration-time curve over 24 hours (AUC24h) and the maximum observed plasma concentration (Cmax)
Toxicity endpoint: termination from treatment due to a suspected adverse drug reaction (SADR) | Measured through Week 24
Toxicity endpoint: adverse events (AEs) or laboratory toxicities of Grade 3 or higher severity judged to be at least possibly attributable to the study medication | Measured through Week 24
Toxicity endpoint: death | Measured through Week 24

SECONDARY OUTCOMES:
AEs or laboratory toxicities of Grade 3 or higher severity judged to be at least possibly attributable to the study medications | Measured through Week 48
Adverse events meeting the International Conference on Harmonisation (ICH) seriousness criteria | Measured through participant's last study visit (through Week 48 or, for participants in long-term safety follow-up, through Week 240)
Treatment discontinued due to toxicity or virologic failure | Measured through participant's last study visit (through Week 48 or, for participants in long-term safety follow-up, through Week 240)
Failure to suppress plasma HIV RNA to less than 400 copies/mL (confirmed within 2 to 4 weeks) | Measured at Week 24 and Week 48
Failure to achieve undetectable plasma HIV RNA (less than 40 copies/mL on Abbott RealTime HIV-1 assay, confirmed within 2 to 4 weeks) | Measured at Week 24 and Week 48
Virologic outcome as per Snapshot and time to loss of virologic response (TLOVR) | Measured at Week 24 and Week 48
Sustained decline in absolute CD4 percent of greater than 5% any time after 12 weeks of therapy | Measured through Week 48
Long-term safety (AEs, toxicities of Grade 3 or higher severity, or deaths at least possibly related to treatment) after 48 weeks | Measured through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Ann Melvin, MD, MPH, Study Chair — Seattle Children's Hospital